CLINICAL TRIAL: NCT05705180
Title: The Influence of Trained Immunity in COVID-19 Vaccinated Individuals
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wuerzburg University Hospital (Other)
Responsible Party: Principal Investigator, Martina Prelog, Prof. Dr., Wuerzburg University Hospital
Other Study IDs: 10.940-3.22_VXSS-218827
Record Dates: First submitted 2023-01-26; First posted 2023-01-30 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Zoster Varicella; Vaccination; Infection
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Serum samples, peripheral blood mononuclear cells (PBMCs)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A Retrospective samples: Retrospective (samples already stored, CoVaKo study cohort): Retrospective samples were consecutively collected during March 2020 and March 2022 (n=420).
  Group 1A: RZV 1-12 months before COVID-19 -mRNA vaccination Group 1B: no RZV (control arm)
  Interventions: Biological: recombinant adjuvanted zoster vaccine
- B Prospective samples: Prospective (samples to be recruited, CoVaKo study cohort): Prospective samples will be collected April 2022 to July 2022 (n=180).
  Group 2A: RZV 1-12 months before COVID-19 -mRNA vaccination Group 2B: no RZV (control arm)
  Interventions: Biological: recombinant adjuvanted zoster vaccine

INTERVENTIONS:
Biological: recombinant adjuvanted zoster vaccine — vaccination with recombinant adjuvantes zoster vaccine

SUMMARY:
The concept of trained immunity defines the long-term functional reprogramming of innate immune cells, which is evoked by exogenous or endogenous insults and leads to an altered response towards a second challenge after return to a non-activated state and is characterized by several markers, such as specific cytokines, activation markers of innate immune cells and epigenetic modifications, e.g. H3K4me3. Vaccinations have been shown to induce trained immunity and to have heterologous effects on other infections or vaccinations. A recent article showed, that individuals who had received recombinant adjuvanted zoster vaccine (RZV) before the pandemic had a 16% lower risk of COVID-19 diagnosis and a 32% lower risk of hospitalization suggesting a protective heterologous effect of RVZ on COVID19 infections. So far, the mechanisms behind these add-on benefits of RZV vaccination are on the hypothetical level and need further experimental evidence.

Therefore, we aim to investigate the specific humoral and cellular immune response towards COVID-19 vaccine in healthy individuals who were exposed to RZV 1 to 12 months before COVID-19 vaccination compared to individuals who did not receive RZV before. Particular emphasis is layed on COVID-19 vaccine non-responders and individuals with breakthrough infections indicating lower vaccine efficacy compared to those who had no breakthrough infection.

The primary objective is the cytokine profile of spike protein-stimulated T, NK and NKT cells. Spike protein stimulated T, NK and NKT cells are characterized by cell surface markers, transcription factor expression, chemokine receptor expression, activation and proliferation markers and by their lineage-specific cytokine pattern. CD14+ monocytes are magnetically isolated and further characterized by cell-culture experiments imitating a training and resting period after stimulation. Epigenetic modifications by methylation of CpG regions are assessed at promoter, enhancer and regulatory gene regions of immune cell characteristic transcription factors by bisulfite conversion and pyrosequencing. Chromatin immunoprecipitation and ChIP-seq will be performed for analysis H3K4me3 associated with trained immunity. Humoral and cellular reactivity to spike protein is analyzed by adapted ELISA and neutralisation assays and by ELISpot and flow cytometry, respectively, and correlated.

From our findings we expect to learn about the role of previous RZV on immunogenicity and efficacy of COVID-19 vaccination and whether mechanisms of trained immunity play a role for better responses towards COVID-19 vaccination.

ELIGIBILITY:
Inclusion Criteria:

Group 1, retrospective (samples already stored, CoVaKo study cohort): healthy (n=420) Group 2, prospective (samples to be recruited, CoVaKo study cohort): healthy (n=180)

* Age 18-90 years, stratified into <60 and ≥60 years
* at least 2 COVID-19-mRNA vaccinations as equivalent to primary immunization and the third and/or fourth dose considered as booster, as recommended for all individuals >12 years (third dose) and for risk groups, medical staff, nursing home residents (fourth dose) in Germany Only individuals naive for SARS-CoV-2 (negative N-specific and S-specific-IgG antibody status, no history of PCR+ swab) before COVID-19 vaccination will be included.

Exclusion Criteria:

* High-dose glucocorticoids >10 mg/day
* Immunosuppressive therapy
* Biologics or immunomodulators
* Transplantation
* Cancer
* Autoimmunity
* RZV after COVID-19 vaccination
* COVID-19 PCR+ before COVID-19 vaccination
* Other types of COVID-19 vaccines than mRNA vaccines

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Immunologically healthy individuals who were vaccinated at least twice with COVID-19 mRNA vaccine (either Comirnaty or Moderna) are taken from CoVaKo study cohort (Group A). Immunologically healthy is defined at inclusion by normal leucocyte and lymphocyte counts, normal CRP and ESR according to age range, no severe allergies requiring daily therapy, no congenital or acquired immunodeficiency or immunosuppression.
  A control group (Group B) consists of individuals who did not receive RZV 1-12 months before COVID-19 vaccination.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Interferon-gamma | 12 months
  Spot forming units in Interferon-gamma ELISpot assay

SECONDARY OUTCOMES:
Spike-specific IgG antibodies | 12 months
  Spike-specific IgG antibodies measured in BAU/ml
Spike-specific IgG antibody avidity | 12 months
  Spike-specific IgG antibody avidity measured in relative avidity by adapted ELISA

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Wuerzburg, Würzburg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No